CLINICAL TRIAL: NCT03639441
Title: Efficacy of Dry Needling for Knee Osteoarthritis: A Single-Blind and Randomized-Controlled Trial
Brief Title: Dry Needling Treatment for Knee Osteoarthritis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Li-Wei Chou, Minister of Rehabilitation, China Medical University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUH107-REC2-100
Record Dates: First submitted 2018-08-16; First posted 2018-08-21 (Actual); Last update posted 2019-08-20 (Actual); Status verified 2018-08

CONDITIONS: Knee Osteoarthritis
Keywords: dry needling; myofascial trigger point; muscle tone
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Dry Needling; Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dry needling (Experimental): In this arm, the subjects will receive the intervention of DN on Day1, Day2 and Day4, in total 3 treatments and will be arrange to take efficacy two assessment on Day8 and Day15, separately.
  Interventions: Procedure: dry needling
- Transcutaneous Electric Nerve Stimulation (Active Comparator): In this arm, the subjects will receive the intervention of Transcutaneous Electric Nerve Stimulation on Day1, Day2 and Day4, in total 3 treatments and will be arrange to take efficacy two assessment on Day8 and Day15, separately.
  Interventions: Procedure: Transcutaneous electrical nerve stimulation

INTERVENTIONS:
Procedure: dry needling — Dry needling, also known as myofascial trigger point dry needling, is an well-proved technique in alternative medicine similar to acupuncture. It involves the use of either solid filiform needles or hollow-core hypodermic needles for therapy of muscle pain, including pain related to myofascial pain syndrome. Dry needling is sometimes also known as intramuscular stimulation (IMS).
  Arms: Dry needling
Procedure: Transcutaneous electrical nerve stimulation — Transcutaneous electrical nerve stimulation (TENS or TNS) is the use of electric current produced by a device to stimulate the nerves for therapeutic purposes.
  TENS, by definition, covers the complete range of transcutaneously applied currents used for nerve excitation although the term is often used with a more restrictive intent, namely to describe the kind of pulses produced by portable stimulators used to treat pain. The unit is usually connected to the skin using two or more electrodes. A typical battery operated TENS unit is able to modulate pulse width, frequency and intensity. Generally TENS is applied at high frequency (>50 Hz) with an intensity below motor contraction (sensory intensity) or low frequency (<10 Hz) with an intensity that produces motor contraction.
  Arms: Transcutaneous Electric Nerve Stimulation

SUMMARY:
The population affected by degenerative knee arthritis is very large. The investigator performed dry needle (DN) treatments with acupuncture needles. This experiment used a randomized single-blind experiment to assess the immediate, short-term and long-term effects of dry needle therapy on patellar pain in patients with degenerative arthritis.

DETAILED DESCRIPTION:
The population affected by degenerative knee arthritis is very large. According to a survey conducted by the Ministry of Health and Welfare, the prevalence of osteoarthritis of the knee in Taiwan is about 3.5 million people, accounting for about 15% of the total population. Its effects are a heavy burden on socio-economic costs, and in addition to being included in medical expenses, serious cases can lead to incapacity to work; therefore, the disease is an important factor in causing disability and disability First, it is worth our attention.

The investigator performed dry needle (DN) treatments with acupuncture needles. Stimulating the effected muscle, the investigator move the needle forward and backward several times. Muscle twitch may occur by our procedure. The pain caused by myofascial trigger points can be decreased effective simultaneously. So far, there is no solid research or clinical trial to evaluate the efficacy of the treatment yet.

For the reasons of the degenerative arthritis pain, the clinical observation is not entirely due to the cause of joint deformity or cartilage damage, soft tissue lesions around the knee is also a common source of pain, the use of dry needle for the diagnosis of soft tissue injury , And observed its efficacy, which is also the core of this study.

This experiment used a randomized single-blind experiment to assess the immediate, short-term and long-term effects of dry needle therapy on patellar pain in patients with degenerative arthritis. The assessment tools included the VAS, WOMAC , Lequesnes index, Gait speed test and the Muscle Tension Changes in the Lower Extremities.

ELIGIBILITY:
Inclusion Criteria:

1. Volunteers who are older than 50 years old and can cooperate with the experiment
2. Established diagnosis of unilateral or bilateral degenerative knee arthritis.
3. There is a local trigger point around the unilateral or bilateral knee joint which on the muscle of Vastus lateralis, Vastus medialis, Gastrocnemius, or Tibialis anterior.

Exclusion Criteria:

1. There are contraindications to general treatment, such as serious medical problems, recent serious trauma, or pregnant women.
2. There has been a history of drug abuse (including excess alcohol) that affects pain assessors.
3. Have received knee surgery.
4. People with central or peripheral nerve disease.
5. Cognitive impairment, unable to cooperate with the experimenter.
6. Patients currently receiving other treatments for knee osteoarthritis

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-02 (Actual); Primary Completion 2019-05-07 (Actual); Study Completion 2019-05-21 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scales | 1 day
  The visual analogue scale or visual analog scale (VAS) is a psychometric response scale which can be used in questionnaires. This tool used to help a person rate the intensity of certain sensations and feelings, such as pain. A straight line of 100mm is actually marked with 0 mm on the far left and 100mm on the far right. Two faces are drawn on both ends. Explain to the patient that 0 mm means no pain and 100 mm means very painful. From the left end The right shift indicates more and more pain. Take a pen and let the patient draw a short line vertically on the line, representing his painful position, and record the measured cm value. In this test, if the score of the subject decreases, it can represent the treatment is helpful for the improvement of the patient's pain.

SECONDARY OUTCOMES:
Pressure Pain Threshold | 1 day
  Pressure pain threshold (PPT) is defined as the minimum force applied which induces pain. This measure has proven to be commonly useful in evaluating tenderness symptom
Muscle tension | 1 day
  Muscle tension is the muscle's resistance to passive stretch during resting state. The measuring tool called Myotone will calculate three parameters such as tone, elasticity and stiffness automatically and get a value to represent the muscle tension. If the value decrease, it can represent the treatment is helpful for the subjective muscle relax.
Gait speed test | 1 day
  The measurement method is to ask the patient to walk a distance of four meters, and then the time taken by the tester to measure, take two measurements and take the average value. In this experiment, the function of the patient's walking is mainly measured by this evaluation method. Whether it is improved, if the patient's walking time is reduced, it can effectively prove the patient's exercise performance.

CONTACTS AND LOCATIONS:
Locations (1):
- China Medical University Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided